CLINICAL TRIAL: NCT01160315
Title: A Prospective Open Randomized Trial on the Efficacy of Gonadotropin-releasing Hormone Agonist Depot-Triptorelin- to Prevent Chemotherapy Induced Premature Ovarian Failure in Lymphoma Patients.
Brief Title: Efficiency of Gonadotropin-releasing Hormone (GnRH) Agonist in Preventing Chemotherapy Induced Ovarian Failure
Acronym: Erasme-POF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ErasmeUH
Record Dates: First submitted 2010-07-07; First posted 2010-07-12 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Fertility Preservation; Alkylating Agents; Lymphoma
Keywords: ovarian failure, chemotherapy, lymphoma, GnRH agonist
MeSH Terms: conditions — Lymphoma | interventions — Triptorelin Pamoate; Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (GnRha arm) (Experimental): IM injection of Triptorelin -Decapeptyl PR 11.25mg- (every 3 months) and Norethisterone acetate- Primolut-Nor 5 mg- per os continuously until the end of the chemotherapy
  Interventions: Drug: Triptorelin; Drug: Norethisterone acetate
- Arm B (control Arm) (Active Comparator): Norethisterone acetate alone, 5mg par day, (ARM B) until the end of the chemotherapy.
  Interventions: Drug: Norethisterone acetate

INTERVENTIONS:
Drug: Triptorelin — Triptorelin: intramusculAR injection every 3 months
  Other Names: Decapeptyl
  Arms: Arm A (GnRha arm)
Drug: Norethisterone acetate — 5 mg/day per os until during chemotherapy
  Other Names: Primolut

SUMMARY:
Chemotherapy drugs like alkylating agents are frequently used in various combined regimens to treat neoplastic and benign diseases. These drugs are definitely associated with premature ovarian failure (POF), resulting in an important decrease of the long-term quality of life and an increase of morbidity. A recent study showed that the patients treated by alkylating agents had a 4.52 fold higher risk to lose their ovarian function compared with those who were treated by other agents. The rate of POF after treatment ranged from 40 to 80%, according to the age of the patients and the total doses administered.

Young women who experience POF have to face with the prospects of infertility and to consider years of hormonal replacement therapy. The possibility of minimizing gonadal damage by administering of protective therapy during chemotherapy represents an attractive option for these patients.

The aim of this study is to evaluate the protective effect on the ovarian function of the gonadotropin-releasing hormone agonist (GnRha) administered concomitantly to alkylating agents. Preliminary data in the literature on animals (rat and monkeys) are promising. Data in human are, however, highly controversial.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 45 years old with lymphoma.
* Menarche >2year
* Subject treated by chemotherapy-induced ovarian failure including alkylant agents (except less than 8 ABVD)
* Presence of both ovaries (ovarian biopsy or hemiovariectomy for cryopreservation before treatment is accepted).
* Ability to give written informed consent

Exclusion Criteria:

* Hormonal-sensible malignancy
* Chemotherapy or radiotherapy before the inclusion in the study
* Pelvic irradiation including the ovaries or TBI
* Pregnancy
* Patient weight above 110 kg
* Anamnesis of thrombo-embolic processes
* Severe hepatic or renal insufficiency
* Systolic blood pressure >15mmHg or diastolic blood pressure > 90mmHg
* Contraindication of IM injection
* Relevant ovarian abnormalities (Functional follicular cyst are tolerated)
* Anamnesis of premature ovarian failure or irregular cycle (repeated amenorrhoea >2 months)
* Dubin-Johnson and Rotor Syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2002-07; Primary Completion 2010-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Premature ovarian failure rate | 5 years
  Primary endpoint is to evaluate the short and long-term efficacy of triptorelin depot plus progestin versus progestin alone to prevent POF induced by chemotherapy treatment. The ovarian function (FSH, E2, Progesterone, and AMH, presence of spontaneous menstrual cycle and pregnancies) will be evaluated every 3 months during the first 6 months after the end of chemotherapy, every 6 months during the next 18 months and once a year during an additional 5 years. All hormonal treatment has to be interrupted 10 days before the blood test.

SECONDARY OUTCOMES:
Impact of the flare-up effect of Triptorelin | 2 years
  The Triptorelin/Norethisterone treatment has to start if possible 10 days before the beginning of the chemotherapy (time necessary to obtain the inhibitory effect of the Gn-Rha on the ovarian function)and at least the same day. The impact of the interval between the triptorelin/noresthisterone treatment and the start of the chemotherapy on the efficacy to protect ovarian function (FSH level at 2 years of follow-up) will be evaluated.
Ovarian function during the treatment | 1 year
  Evaluation of the inhibitory action of the treatment on ovarian function during the chemotherapy: the hormonal profile (FSH and estradiol levels) will be evaluated 10 days after the triptorelin/Norethisterone treatment start, before the second injection (3 months) and at the end of the chemotherapy. Adverse effects due to the injection are evaluated 7-10 days after each injection.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year
  Anamnesis including the compliance of the treatment (possible treatment interruption or dosage modification) and the adverse events are performed at each visit. All events expected and directly related to the chemotherapy or the initial pathology will be documented in the Case Report Form adverse events. Specific anamnesis concerning the possible adverse events due to treatment must be completed for each follow-up visit.
Add back therapy effect | 1 year
  Evaluation of the efficacy of concomitant administration of progestin alone as "Add Back Therapy" during the treatment: specific anamnesis including estrogen-deficiency symptoms (hot flushes, vaginal dryness...) is reported at each visit during the treatment. Osteodensitometry is performed after 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Englert, MD, PhD, Study Director — Erasme University Hospital
Locations (15):
- Belgium (7):
  - Algemeen Ziekenhuis Stuivenberg, Antwerp
  - AZ St Jan, Brugges
  - Bordet, Brussels
  - Erasme Hospital, Brussels
  - AZ-VUB, Brussels
  - St Luc University, Brussels
  - CHRU Lille, Lille
- France (7):
  - CHU Dijon, Dijon
  - CHU Nancy, Nancy
  - Hôpital Hotel Dieu, Paris
  - St Louis Hospital, Paris
  - CHU St Antoine, Paris
  - Henry-Mondor Hospital, Paris-Creteil
  - Centre Henri Beckerel, Rouen
- Instituto Europeo di oncologia, Milan, Italy

REFERENCES:
- [Derived] Demeestere I, Brice P, Peccatori FA, Kentos A, Gaillard I, Zachee P, Casasnovas RO, Van Den Neste E, Dechene J, De Maertelaer V, Bron D, Englert Y. Gonadotropin-releasing hormone agonist for the prevention of chemotherapy-induced ovarian failure in patients with lymphoma: 1-year follow-up of a prospective randomized trial. J Clin Oncol. 2013 Mar 1;31(7):903-9. doi: 10.1200/JCO.2012.42.8185. Epub 2012 Nov 5. PMID 23129737